CLINICAL TRIAL: NCT02381340
Title: Effect of the BaroSense ACE Stapler Procedure on Food Intake, Food Reward, Gastric Emptying, Hormone Release, Inflammatory Profile, Gut Microbiota and Behaviour Towards Food.
Brief Title: ACE Stapler Sub Study
Status: Completed | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Boston Scientific Corporation (Industry); BaroSense Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: NL39402.068.12
Record Dates: First submitted 2015-03-02; First posted 2015-03-06 (Estimated); Last update posted 2018-01-12 (Actual); Status verified 2015-03

CONDITIONS: Obesity
Keywords: Obesity; Bariatric surgery; Gastric plication; Minimal invasive surgery; gastrointestinal hormones; food-reward; satiety; microbiota
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma samples, faeces
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: ACE stapling procedure — Endoscopic trans-oral gastroplication

SUMMARY:
Obesity and its associated conditions have reached epidemic proportions. Estimates are that about one third of the adults in the United States have obesity. At this moment there are many therapeutic approaches for the treatment of obesity. But, efficacy of most treatment options are limited and so far surgical intervention has been proven to be the only strategy to overcome severe obesity. However, bariatric surgery has limitations and risks, which might be minimized by non-incisional endoscopic procedures.

BaroSense developed a new device, called the Articulating Circular Endoscopic (ACETM) Stapler, which can be used in the treatment of obesity. It is a trans-oral procedure, which intends to reduce the ability of the stomach to expand by creating plications in the region of the fundus and greater curvature. In contrast with other bariatric surgery it is endoscopically performed, reversible and if it fails most future surgical options are still open.

The main study ('Open, prospective study to evaluate the safety and preliminary effectiveness of the BaroSense ACE™ Stapler for the treatment of obesity', multicenter study (MUMC+, AMC and St. Antonius), accepted by MEC AMC) seeks to determine the safety and efficacy of this plicating system for patients with severe obesity.

In this sub-study the investogators want to unravel the exact mechanism and provide more information about the efficacy of the BaroSense ACE™ Stapler. Therefore the authors will measure changes in various parameters that are known to affect weight loss and metabolism, before and after gastric plication (by using the BaroSense ACE™ Stapler) in overweight subjects (these parameters will only be measured in patients at MUMC+). These parameters are post-prandial satiety, food-reward and related brain signalling, gastric emptying, behaviour towards food, food intake, satiety hormone release, microbiota composition and inflammatory markers.

Objectives:

Aim of the present study will be to assess the effect of the BaroSense ACE™ stapler on postprandial satiety, food-reward and related brain signalling, gastric emptying, behaviour towards food, food intake, hormone release, microbiota composition and inflammatory markers.

ELIGIBILITY:
Inclusion Criteria:

Criteria for inclusion in main ACE stapling study:

* Subject must be able to understand and be willing to sign an informed consent document.
* Subject must be willing and able to participate in all aspects of the study and agree to comply with all study requirements for the duration of the study. This includes availability of reliable transportation and sufficient time to attend all follow-up visits.
* Subject has a BMI of 40 - 45 or 30 to 39.9 plus one or more co-morbid diseases expected to improve with weight loss, including but not limited to hypertension, dyslipidemia, obstructive sleep apnea, or diabetes mellitus.
* Subject must be fully ambulatory, without chronic reliance on walking aids such as crutches, walkers or a wheelchair.
* Subject must be of sufficient and stable medical health, as evaluated by the Principal Investigator.
* Subject must have a primary care physician that will manage the subject for any co-morbid conditions throughout the study.
* Subject must have failed standard obesity therapy of diet, exercise, behaviour modification, and pharmacologic agents either alone or in combination, as assessed by an interview with a member of the study team at baseline.
* Subject agrees to refrain from any type of reconstructive surgery that may affect body weight such as mammoplasty or abdominal lipoplasty or liposuction, during the trial.

Inclusion criteria sub study

• Patient must be included in the main study

Exclusion Criteria:

Main study

* Subject has history of/or signs and/or symptoms of gastro-duodenal ulcer disease.
* Subject has poorly controlled diabetes as indicated by the lack of stable diabetes medications and doses over the last month, or has a history of diabetes for greater than 10 years.
* Subject has had significant weight loss in the last 3 months, or between baseline and the study procedure.
* Subject has a history or is diagnosed with eating disorders.
* Subject has history of peptic ulcer and tests positive for H. pylori, unless treated before the procedure.
* Subject has symptomatic congestive heart failure, cardiac arrhythmia or unstable coronary artery disease.
* Subject has pre-existing respiratory disease such as chronic obstructive pulmonary disease (COPD), pneumonia or cancer.
* Subject has significant esophageal disease including Zenker's diverticulum, grade 3-4 reflux esophagitis, stricture, Barrett's esophagus, esophageal cancer, esophageal diverticulum, dysphagia, achalasia, or symptoms of dysmotility.
* Subject is observed during EGD to have heavily scarred, malignant or poor quality/friable tissue in areas of the stomach where plications are to be placed.
* Subject has renal and/or hepatic insufficiency.
* Subject has thyroid disease which is not controlled with medication.
* Subject has a history of intestinal strictures or adhesions.
* Subject has systemic infection in the body at the time of the plication procedure.
* Female subject who is pregnant (i.e., has a positive urine or blood pregnancy test prior to the procedure), is suspected to be pregnant, is lactating or is of childbearing potential but refuses to use adequate contraception during the study.
* Female subject who started birth control pills less than 3 months before enrollment, or who plans to start taking birth control pills during the study.
* Subject has had previous bariatric, gastric or esophageal surgery; intestinal obstruction; portal gastropathy; gastrointestinal tumors; esophageal or gastric varices, or gastroparesis.
* Subject has severe coagulopathy (prothrombin time > 3 seconds over control or platelet count < 100,000) or is presently taking heparin, coumadin, warfarin, or other anticoagulants or other medications which impede coagulation or platelet aggregation.
* Subject has chronic/acute upper GI bleeding conditions.
* Subjects who are unable to discontinue use of aspirin and/or non-steroidal anti-inflammatory agents (NSAIDs) at least 14 days prior to a plication procedure and continuing for 14 days post-procedure.
* Subjects undergoing chronic steroid therapy.
* Subjects undergoing immunosuppressive therapy.
* Subjects who cannot discontinue either prescription or over the counter weight loss medications for at least 30 days prior to the procedure as well as during the trial period.
* Subjects who have started medications within the last 3 months that are known to cause weight gain.
* Subjects who have cardiac pacemakers or other electronic implantable devices.
* Subjects who have hiatal hernias greater than 2 cm.
* Subjects who have current or potential neck masses that in the opinion of the investigator, may interfere with study-related procedures, or has a Mallampati (intubation) score greater than 3.
* Subjects who have poorly controlled psychiatric disease including but not limited to manic-depressive disorder, schizophrenia, borderline personality disorder, depression or suicidal tendencies.
* Subject has Crohn's disease or Ulcerative Colitis.
* Subject currently uses or has a history of illicit drug(s) or abuses alcohol (defined as regular or daily consumption of more than 4 alcoholic drinks per day).
* Subject has participated in a clinical study with an investigational new drug, biological, or therapeutic device within ≤ 28 days prior to enrollment in this study, and does not agree to abstain from participation in other clinical trials of any kind during this study.

Exclusion criteria sub study

* Presence of contra-indications for MRI and f-MRI, as mentioned in Attachment 1 and 2.
* Hypersensibility to contrast (Dotarem)
* Claustrophobia
* Pregnancy

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients that will undergo an ACE stapling procedure for the treatment of obesity.
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2012-06; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Satiety, food intake and hunger | 1 year
  This will be evaluated in a test day before, 1 month after and 12 months after the procedure

SECONDARY OUTCOMES:
Changes in gastrointestinal hormone release | 1 year
  GLP-1, PYY and ghrelin
Gastric emptying | 1 year
  Evaluated with 13C octanoic acid breath test and real-time MRI
Behavior towards food and brain-related signaling | 1 year
  Evaluated with fMRI, questionnaires (eating behavior) and computer tasks (liking, wanting)
Inflammatory status | 1 year
  By evaluating inflammatory plasma markers

CONTACTS AND LOCATIONS:
Locations (1):
- Maastricht University Medical Center, Maastricht, Limburg, Netherlands

REFERENCES:
- [Derived] Paulus GF, van Avesaat M, Crijnen JAW, Ernest van Heurn LW, Westerterp-Plantenga MS, Bouvy ND. Preliminary evidence that endoscopic gastroplication reduces food reward. Appetite. 2020 Jul 1;150:104632. doi: 10.1016/j.appet.2020.104632. Epub 2020 Feb 15. PMID 32070711